CLINICAL TRIAL: NCT00679627
Title: A Randomized, Double-Blind, Placebo-controlled Trial of Long-term (2-year) Treatment of Galantamine in Mild to Moderately-Severe Alzheimer's Disease
Brief Title: A Study of Galantamine Used to Treat Patients With Mild to Moderate Alzheimer's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to a pre-specified imbalance of deaths between treatment groups, the DSMB recommended early termination of the trial
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR012463; GALALZ3005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Results first posted 2013-09-02 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Galantamine; Dementia, Alzheimer type; Memory loss
MeSH Terms: conditions — Alzheimer Disease; Memory Disorders | interventions — Galantamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Galantamine (Experimental): Galantamine 8mg/ day oral capsule increased to 16mg/day then to 24 mg per day
  Interventions: Drug: Galantamine
- Placebo (Placebo Comparator): Matching placeco
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Galantamine — 8mg/ day oral capsule increased to 16mg/day then to 24 mg per day
  Arms: Galantamine
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of 2 years of treatment with galantamine as compared with placebo of patients who have mild to moderately severe Alzheimer's disease (AD).

DETAILED DESCRIPTION:
This is a long-term (2-year), randomized (patients will be assigned to treatment by chance), double blind (neither the physician nor the patient will know which treatment is assigned) study of galantamine versus placebo in subjects with mild to moderately-severe AD. Approximately 2,000 patients will participate in this study. The study length for each patient is approximately 25.5 months. The study consists of 3 phases: a pretreatment phase, a treatment phase, and a posttreatment phase. The pretreatment phase includes a 2-week screening period (to obtain a patient's and his or her caregiver's informed consent and to confirm eligibility for the study) and a baseline visit at which subjects will be randomly assigned, in a 1 to 1 ratio, to receive either galantamine or placebo once a day in the morning. Study drug will first be dispensed at the baseline visit. The treatment phase is composed of a titration period (the study drug will be introduced gradually) and a maintenance period and includes 9 visits (3 of which are conducted by telephone). The titration period is 12 weeks long, and visits occur about every 28 days. In the first 4 weeks of the titration period, subjects will receive either 8 mg galantamine or matching placebo, and this dose will be increased to 16 mg galantamine or placebo in the second 4 weeks. The dose will then be increased to 24 mg galantamine or placebo for the final 4 weeks of the titration period if the investigator believes the subject will benefit from and will safely tolerate 24 mg/day. If not, the subject may continue to receive 16 mg galantamine or placebo through the end of the titration period. After the titration period, subjects will enter the maintenance period and continue to take study drug at the dosage they received at the end of the titration period. This dosage may be continued through the end of the study or may be changed once (either up from 16 to 24 mg or down from 24 to 16 mg), depending upon the benefit and the safety of such a change for the individual patient as judged by the investigator. No dosage will exceed 24 mg/day. The posttreatment phase includes an End-of-Study Visit that occurs at the end of the maintenance period. A follow-up telephone contact (interview) is conducted 1 month after the End-of-Study Visit. The effectiveness of galantamine will be evaluated using the following tools: the Mini-Mental State Examination (MMSE); the Disability Assessment in Dementia (DAD); and the Assessment of Patient Accommodation Status and Caregiver Burden (APAS CarB). Safety evaluations for the study include the monitoring of vital status and institutionalization status, adverse events, vital signs, weight, physical and neurologic examinations. A Data Safety Monitoring Board, external to the company, has been commissioned for this study to monitor the progress of the study and to ensure that the safety of patients is not compromised. The effectiveness hypothesis of this study is that galantamine, 16 to 24 mg per day, is superior to placebo in reducing cognitive decline from baseline (start of study drug) as measured by the MMSE over the course of 2 years. The safety hypothesis is that the mortality rate in the galantamine 16 to 24 mg per day treatment group will be the same as that in the placebo group over the course of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* diagnosed with mild to moderately-severe, probable or possible AD, established in accordance with the criteria defined by the National Institute of Neurological and Communicative Disorders and Stroke and Alzheimer's Disease Related Disorders Association or the Diagnostic and Statistical Manual, Fourth Edition
* living with or have regular and frequent visits from a responsible caregiver.

Exclusion Criteria:

* Neurodegenerative disorders other than AD, such as Parkinson's Disease, Frontotemporal Dementia or Huntington's disease
* Any of specified conditions which may contribute to dementia
* any of specified coexisting diseases, including significant cardiovascular disease.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2051 (Actual)
Dates: Start 2008-06; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (95):
- Czechia (5):
  - Hradec Králové
  - Mìlník 1
  - Olomouc
  - Ostrava
  - Prague
- Estonia (4):
  - Tallinn
  - Tartu
  - Viljandi
  - Vorumaa
- Limoges, France
- Germany (26):
  - Bad Aibling
  - Bad Homburg
  - Bad Honnef
  - Bamberg
  - Berlin
  - Bielefeld
  - Bochum
  - Butzbach
  - Franfurt
  - Fürth
  - Gelsenkirchen
  - Göttingen
  - Hamburg
  - Hanover
  - Hattingen
  - Karlstadt am Main
  - Leverkusen
  - Lüneburg
  - Mittweida
  - Mönchengladbach
  - Nuremberg
  - Oldenburg
  - Ulm
  - Unterhaching
  - Westerstede
  - Wiesbaden
- Greece (3):
  - Athens
  - Heraklion Crete
  - Thessalonikis
- Riga, Latvia
- Lithuania (3):
  - Kaunas
  - Šiauliai
  - Vilnius
- Romania (8):
  - Arad
  - Bucharest
  - Bucharest Sector 5
  - Cluj-Napoca
  - Constanța
  - Craiova
  - Iași
  - Tg Mures
- Russia (19):
  - Kazan'
  - Kazan’
  - Kirov
  - Krasnodar
  - Lipetsk
  - Moscow
  - Moscow Russia
  - Nizny Novgorod
  - Novosibirsk
  - Rostov-on-Don
  - Saint Petersburg
  - Samara
  - Saratov
  - Smolensk
  - Smolensk Region N/A
  - Tomsk Na
  - Voronezh
  - Yaroslavl
  - Yekaterinburg
- Slovakia (7):
  - Bratislava
  - Dubnica nad Váhom
  - Košice
  - Plešivec
  - Spišská Nová Ves
  - Šenkvice
  - Vranov nad Topľou
- Slovenia (4):
  - Kamnik
  - Lesce
  - Ljubljana
  - Maribor
- Ukraine (14):
  - Chernivtsy
  - Dnipro
  - Dnipropetrovsk
  - Donetsk
  - Kharkiv
  - Kherson
  - Kiev
  - Kyiv
  - Lviv
  - Odesa
  - Poltava
  - Simferopol
  - Uzhhorod
  - Vinnitsa

REFERENCES:
- [Derived] Lim AWY, Schneider L, Loy C. Galantamine for dementia due to Alzheimer's disease and mild cognitive impairment. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD001747. doi: 10.1002/14651858.CD001747.pub4. PMID 39498781
- [Derived] Hager K, Baseman AS, Nye JS, Brashear HR, Han J, Sano M, Davis B, Richards HM. Effect of concomitant use of memantine on mortality and efficacy outcomes of galantamine-treated patients with Alzheimer's disease: post-hoc analysis of a randomized placebo-controlled study. Alzheimers Res Ther. 2016 Nov 15;8(1):47. doi: 10.1186/s13195-016-0214-x. PMID 27846868
- [Derived] Hager K, Baseman AS, Nye JS, Brashear HR, Han J, Sano M, Davis B, Richards HM. Effects of galantamine in a 2-year, randomized, placebo-controlled study in Alzheimer's disease. Neuropsychiatr Dis Treat. 2014 Feb 21;10:391-401. doi: 10.2147/NDT.S57909. eCollection 2014. PMID 24591834

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study investigated the benefits and risks of long-term galantamine use in participants with Alzheimer's Disease. The study was conducted from 19 May 2008 to 20 May 2012 at 127 clinical centers in 13 countries. A total of 2051 participants were randomized to study treatment, of these 2045 received at least 1 dose of treatment.
Pre-assignment Details: The Data Safety Monitoring Board (DSMB) recommended that the study be terminated early because of an imbalance of deaths between the treatment groups.
Groups:
- Placebo: During the titration and long-term maintenance periods, placebo was supplied as oral capsules matching galantamine capsules in size and appearance. The study drug was administered using the same titration and maintenance regimens as was used for participants in the galantamine treatment group.
- Galantamine: During the titration period (Days 1 to 84), participants received galantamine controlled-release oral capsules 8 mg/day for the first 4 weeks, followed by 16 mg/day for the next 4 weeks, then 24 mg/day for the next 4 weeks (based on tolerability). During the long-term maintenance period (Months 4 to 24), participants received galantamine at the dosage achieved at Day 84 of the titration period and continued until the completion of the Month 24 visit. A one-time dose titration to 16 or 24 mg/day was allowed, based on the investigator's judgment and participant tolerability.
Period: Overall Study
Arm/Group | Placebo | Galantamine
Started | 1021 | 1024
Completed | 322 | 339
Not Completed | 699 | 685
Not completed — Death | 41 | 29
Not completed — Adverse Event | 43 | 53
Not completed — Withdrawal by Subject | 168 | 172
Not completed — Lost to Follow-up | 22 | 26
Not completed — Early Study Closure | 425 | 405

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Galantamine | Total
Number analyzed (Participants) | 1021 | 1024 | 2045
Age Continuous [Mean (Standard Deviation); unit: participants] | 73.2 (8.67) | 73 (8.88) | 73.1 (8.77)
Age, Customized [Number; unit: participants]
  <61 | 112 | 112 | 224
  61-<76 | 467 | 466 | 933
  >=76 | 442 | 446 | 888
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 654 | 671 | 1325
  Male | 367 | 353 | 720
Region of Enrollment [Number; unit: participants]
  Czech Republic | 33 | 34 | 67
  Estonia | 53 | 51 | 104
  France | 10 | 11 | 21
  Germany | 218 | 221 | 439
  Greece | 35 | 36 | 71
  Italy | 25 | 24 | 49
  Latvia | 2 | 2 | 4
  Lithuania | 23 | 21 | 44
  Romania | 84 | 84 | 168
  Russia | 274 | 271 | 545
  Slovakia | 85 | 88 | 173
  Slovenia | 13 | 13 | 26
  Ukraine | 166 | 168 | 334

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Mini-Mental State Examination (MMSE) Score
Description: The MMSE is a brief 30-point questionnaire test that is used or the assessment of dementia patients' cognitive impairment. Evaluation of points are as follows: 24 to 30 = no cognitive impairment, 18 to 23 = mild cognitive impairment, 0 to 17 = severe cognitive impairment. Lower scores indicate worsening.
Time Frame: Baseline, Month 24
Population: An intent-to-treat (ITT) with last observation carried forward (LOCF) approach was used for the primary analysis. The ITT analysis set included all randomized participants who received at least 1 dose of treatment and had at least 1 postbaseline MMSE measure.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 906 | 906
Scores on scale | -2.14 (4.340) | -1.41 (4.050)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; Test type: Superiority or Other; p < 0.001, ANCOVA

2. Primary Outcome: The Number of Deaths Reported in Participants
Description: An external Data Safety Monitoring Board (DSMB) was assigned for this study to monitor the progress of the study and to ensure that the safety of participants was not compromised.
Time Frame: Up to 2 years
Population: The safety analysis was performed on the safety population, ie, all randomized participants who received at least one dose of the study drug.
Measure: Number; unit: Number of Participants
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 1021 | 1024
Number of Participants | 56 | 33
Statistical Analysis 1: Comparison: Placebo vs Galantamine; Test type: Superiority or Other; p = 0.011, Regression, Cox; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.37 to 0.89]

3. Secondary Outcome: Change From Baseline in the Mini-Mental State Examination (MMSE) Score
Description: as for outcome 1
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 906 | 906
Scores on scale | -0.28 (2.938) | 0.15 (2.725)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; Test type: Superiority or Other; p < 0.001, ANCOVA

4. Secondary Outcome: Change From Baseline in Disability Assessment in Dementia (DAD) Scores
Description: The DAD assesses physical activities of daily living and instrumental-activities of daily livings of participants with Alzheimer disease. This measure is a validated, disability assessment scale that collects information regarding the ability of a participant to initiate, plan, organize, and perform activities of daily living, as based on a structured interview with the caregiver. The maximum scores were 13 for initiation, 10 for planning and organizing, and 17 for effective performance in order to yield a total maximum score of 40. These scores were normalized to a scale of 100 for analysis.A higher score, or percentage of items that can be performed represents fewer disabilities in carrying out activities of daily living while a lower percentage indicates an increase in disabilities.
Time Frame: Baseline, Month 24
Population: An intent-to-treat (ITT) with last observation carried forward (LOCF) approach was used for the analysis. The ITT analysis set included all randomized participants who received at least 1 dose of treatment and had at least 1 postbaseline DAD measure.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 906 | 906
Scores on scale | -10.81 (18.268) | -8.16 (17.251)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; Test type: Superiority or Other; p = 0.002, ANCOVA

5. Secondary Outcome: Change From Baseline in Patient Accommodation Measured Using the Assessment of Subject Accommodation Status and Caregiver Burden (APAS-CarB)
Description: The APAS-CarB is a measure used to evaluate participant status and caregiver burden. The table below presents Patient Accommodation assessed as the percentage of participants "home with friend or relative" using the APAS-CarB.
Time Frame: Baseline, Months 12 and 24
Population: An intent-to-treat (ITT) with last observation carried forward (LOCF) approach was used for the analysis. The ITT analysis set included all randomized participants who received at least 1 dose of treatment and had at least 1 postbaseline APAS-CarB measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 906 | 906
Percentage of participants
  Home with friend or relative - Baseline | 62.1 | 62.8
  Home with friend or relative - Month 12 | 61.4 | 61.8
  Home with friend or relative - Month 24 | 55.3 | 60.1

6. Secondary Outcome: Change From Baseline in Caregiver Time Spent With the Patient Measured Using the Assessment of Subject Accommodation Status and Caregiver Burden (APAS-CarB)
Description: The table below presents the number of days that caregiving activities were provided during the past week.
Time Frame: Baseline, Months 12 and 24
Population: The ITT analysis set included all randomized participants who received at least 1 dose of treatment and had at least 1 postbaseline measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 906 | 906
Days
  Provided caregiving during past week - Baseline | 5.91 (2.094) | 5.77 (2.241)
  Provided caregiving during past week - Month 12 | 6.06 (1.964) | 6.07 (1.969)
  Provided caregiving during past week - Month 24 | 6.13 (1.952) | 6.20 (1.830)

7. Secondary Outcome: Change From Baseline in Institutional Status
Description: This table describes the number of participants who were reported as institutionalized at baseline and Month 24.
Time Frame: Baseline, Month 24
Population: as for outcome 6
Measure: Number; unit: Number of Participants
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 906 | 906
Number of Participants
  Baseline | 1 | 0
  Month 24 | 5 | 6
Statistical Analysis 1: Comparison: Placebo vs Galantamine; Test type: Superiority or Other; p = 0.269, Cochran-Mantel-Haenszel — Baseline
Statistical Analysis 2: Comparison: Placebo vs Galantamine; Test type: Superiority or Other; p = 0.835, Cochran-Mantel-Haenszel — Month 24

8. Secondary Outcome: Change From Baseline in the Mini-Mental State Examination (MMSE) Subscales (Orientation, Registration, Attention and Calculation, Recall, and Language)
Description: The MMSE, is a validated, brief examination that rates subjects on orientation (total score, 10), registration (total score, 3), attention (total score, 5), calculation (total score, 5), recall (total score, 3), and language (total score, 9). The maximum score is 30 (only the higher of the two scores for attention and calculation [each with a maximum score of 5] was used). A higher score compared with baseline indicates less impairment.
Time Frame: Baseline, Month 24
Population: The ITT analysis set included all randomized participants who received at least 1 dose of treatment and had at least 1 postbaseline MMSE measure.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 906 | 906
Scores on scale
  Orientation | -0.96 (2.320) | -0.76 (2.128)
  Registration | -0.20 (0.771) | -0.16 (0.692)
  Attention and Calculation | -0.46 (1.526) | -0.16 (1.561)
  Recall | 0.00 (1.013) | 0.10 (1.070)
  Language | -0.93 (1.895) | -0.68 (1.867)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; Test type: Superiority or Other; p = 0.194, ANCOVA — Orientation subscale
Statistical Analysis 2: Comparison: Placebo vs Galantamine; Test type: Superiority or Other; p = 0.353, ANCOVA — Registration subscale
Statistical Analysis 3: Comparison: Placebo vs Galantamine; Test type: Superiority or Other; p = 0.009, ANCOVA — Attention and Calculation subscale
Statistical Analysis 4: Comparison: Placebo vs Galantamine; Test type: Superiority or Other; p = 0.158, ANCOVA — Recall subscale
Statistical Analysis 5: Comparison: Placebo vs Galantamine; Test type: Superiority or Other; p = 0.088, ANCOVA — Language subscale

9. Secondary Outcome: Change From Baseline in the Disability Assessment in Dementia (DAD) Subscales (Initiation, Planning and Organization, Effective Performance, Basic, Instrumental, and Leisure)
Description: as for outcome 4
Time Frame: Baseline, Month 24
Population: This analysis was performed in the intent-to-treat population which included all randomized participants who had at least 1 postbaseline DAD measure.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 906 | 906
Scores on scale
  Initiation | -13.53 (22.993) | -9.60 (20.660)
  Planning and Organization | -13.14 (24.565) | -9.96 (23.154)
  Effective Performance | -13.82 (21.975) | -10.82 (19.959)
  Basic | -14.24 (24.093) | -9.84 (21.899)
  Instrumental | -13.52 (23.210) | -10.72 (21.714)
  Leisure | -13.02 (35.370) | -10.46 (32.769)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; Test type: Superiority or Other; p = 0.010, ANCOVA — Initiation subscale
Statistical Analysis 2: Comparison: Placebo vs Galantamine; Test type: Superiority or Other; p = 0.043, ANCOVA — Planning and Organization subscale
Statistical Analysis 3: Comparison: Placebo vs Galantamine; Test type: Superiority or Other; p = 0.018, ANCOVA — Effective Performance subscale
Statistical Analysis 4: Comparison: Placebo vs Galantamine; Test type: Superiority or Other; p = 0.005, ANCOVA — Basic subscale
Statistical Analysis 5: Comparison: Placebo vs Galantamine; Test type: Superiority or Other; p = 0.054, ANCOVA — Instrumental subscale
Statistical Analysis 6: Comparison: Placebo vs Galantamine; Test type: Superiority or Other; p = 0.137, ANCOVA — Leisure subscale

ADVERSE EVENTS:
Time Frame: Over 2 years
Arm/Group | Placebo | Galantamine
Serious Adverse Events (participants affected / at risk) | 123/1021 | 129/1024
Other Adverse Events (participants affected / at risk) | 115/1021 | 168/1024
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1021) | Galantamine (N=1024)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 3 | 10
Cardiac Failure Acute (Cardiac disorders) | 2 | 2
Cardio-Respiratory Arrest (Cardiac disorders) | 3 | 0
Cardiopulmonary Failure (Cardiac disorders) | 4 | 3
Cardiovascular Insufficiency (Cardiac disorders) | 3 | 1
Ischaemic Cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 2 | 6
Myocardial Ischaemia (Cardiac disorders) | 1 | 1
Postinfarction Angina (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 2
Cataract Subcapsular (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 2
Lens Disorder (Eye disorders) | 0 | 1
Anal Polyp (Gastrointestinal disorders) | 1 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Enterocolitis Haemorrhagic (Gastrointestinal disorders) | 0 | 1
Faecal Incontinence (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 2
Haemorrhagic Erosive Gastritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 2
Intestinal Stenosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophageal Achalasia (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Peritoneal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Varices Oesophageal (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Abasia (General disorders) | 0 | 1
Death (General disorders) | 1 | 0
Hypothermia (General disorders) | 2 | 0
Inflammation (General disorders) | 1 | 0
Multi-Organ Failure (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Sudden Death (General disorders) | 3 | 1
Bile Duct Stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 2
Abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2
Bronchopneumonia (Infections and infestations) | 3 | 2
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0
Ear Infection (Infections and infestations) | 0 | 1
Gastroenteritis Rotavirus (Infections and infestations) | 1 | 0
Gastrointestinal Infection (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 1 | 2
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 8
Post Procedural Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 0 | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0
Carbon Monoxide Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Chemical Poisoning (Injury, poisoning and procedural complications) | 0 | 1
Exposure to Toxic Agent (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 2
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 3 | 2
Femur Fracture (Injury, poisoning and procedural complications) | 3 | 3
Forearm Fracture (Injury, poisoning and procedural complications) | 1 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 2 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 3 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 2
Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 2
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple Fractures (Injury, poisoning and procedural complications) | 1 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Skeletal Injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Urethral Injury (Injury, poisoning and procedural complications) | 0 | 1
Wound Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Blood Pressure Increased (Investigations) | 0 | 1
Weight Decreased (Investigations) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 4
Diabetes Mellitus (Metabolism and nutrition disorders) | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral Disc Compression (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pharyngeal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary Gland Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered State of Consciousness (Nervous system disorders) | 1 | 0
Cerebral Arteriosclerosis (Nervous system disorders) | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 1 | 1
Cerebral Infarction (Nervous system disorders) | 2 | 1
Cerebrovascular Accident (Nervous system disorders) | 2 | 4
Cerebrovascular Disorder (Nervous system disorders) | 1 | 1
Coma (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 2 | 0
Dementia Alzheimer's Type (Nervous system disorders) | 12 | 9
Diabetic Neuropathy (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 3 | 0
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0
Haemorrhagic Stroke (Nervous system disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 8 | 2
Loss of Consciousness (Nervous system disorders) | 1 | 3
Polyneuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Speech Disorder (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 3
Transient Ischaemic Attack (Nervous system disorders) | 3 | 2
Vertebrobasilar Insufficiency (Nervous system disorders) | 0 | 1
Abnormal Behaviour (Psychiatric disorders) | 1 | 0
Adjustment Disorder (Psychiatric disorders) | 0 | 1
Aggression (Psychiatric disorders) | 1 | 3
Agitation (Psychiatric disorders) | 2 | 1
Catatonia (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 0 | 2
Restlessness (Psychiatric disorders) | 1 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 1
Incontinence (Renal and urinary disorders) | 1 | 0
Nephritis (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 1
Renal Failure Chronic (Renal and urinary disorders) | 1 | 0
Stress Urinary Incontinence (Renal and urinary disorders) | 0 | 1
Tubulointerstitial Nephritis (Renal and urinary disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 2
Pelvic Pain (Reproductive system and breast disorders) | 0 | 1
Scrotal Disorder (Reproductive system and breast disorders) | 1 | 0
Vulval Leukoplakia (Reproductive system and breast disorders) | 1 | 0
Acute Lung Injury (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Carotid Artery Stent Removal (Surgical and medical procedures) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
Circulatory Collapse (Vascular disorders) | 1 | 0
Essential Hypertension (Vascular disorders) | 0 | 2
Haemorrhagic Infarction (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypertensive Crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Malignant Hypertension (Vascular disorders) | 1 | 1
Pallor (Vascular disorders) | 1 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1021) | Galantamine (N=1024)
Vertigo (Ear and labyrinth disorders) | 48 | 57
Nausea (Gastrointestinal disorders) | 24 | 85
Headache (Nervous system disorders) | 58 | 58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.